CLINICAL TRIAL: NCT04759690
Title: Effects of Action Observation Training Combined With Exercises on Balance and Risk of Fall Over 65 Years Old
Brief Title: Effects of Action Observation Training and Exercises Over 65 Years Old
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul Medipol University Hospital (Other)
Responsible Party: Principal Investigator, bagdattekkus, Principal Investigator, physiotherapist, Istanbul Medipol University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: p3957ghb
Record Dates: First submitted 2020-12-06; First posted 2021-02-18 (Actual); Last update posted 2022-05-02 (Actual); Status verified 2022-04

CONDITIONS: Fall Prevention; Elderly
Keywords: Aging; Action observation; Balance exercise; Fall prevention

STUDY DESIGN:
Intervention Model Description: Cross-sectional sampling / Randomized controlled trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Action observation and exercise group (Experimental): Action observation group consist of 30 randomly selected participants.Action observation + conventional balance exercise group
  Interventions: Behavioral: Action observation; Behavioral: Exercise group
- Exercise group (Other): Exercise group is the control group.Consist of 30 randomly selected participants. The participants will only do the conventional balance exercise.
  Interventions: Behavioral: Exercise group

INTERVENTIONS:
Behavioral: Action observation — Action observation group: The participants will first watch the conventional balance exercises with the action observation method on video for 15 minutes.After watching of conventional balance exercise for 45 minutes in 5-10 repetitions.
  Other Names: Conventional balance exercises
  Arms: Action observation and exercise group
Behavioral: Exercise group — Exercise group is the control group.TheParticipants will only do the conventional balance exercise without action observation for 45 minutes in 5-10 repetitions.

SUMMARY:
With aging, the decrease in muscle strength in the musculoskeletal system , body biomechanics and posture changes and the risk of falling increase. The greatest danger of falling in this population is risky and the other danger is that it causes fractures, creates physical and psychological trauma, and increases the need for long-term care and health services. Increasing exercise efficiency for balance and preventing falls are extremely important for physical and cognitive health.

İn recent years ,the''Action Observation''approach has been used as an added method to treatments to increase the effectiveness of exercise.Action observation ; it is a cognitive training that triggers motor learning by observing the desired activity and positively affects learning.

The aim of the study : To investigate the effects of exercises on balance and fall risk together with action observation in individuals over 65 years of age . The researchers planned to combine action observation and traditional balance exercises as a group training and compare them with the control group .

The hypothesis of the research is that action observation(AO) will be more useful in maintaining balance and preventing the risk of falling.

Materials and methods of the research:Participants will consist of volunteers over 65 years of age(65-80 years old ). 60 participants to be selected randomly. The participants will be randomly assigned 2 groups.

Experimental group :( 30 participants ) Action observation+ exercise combination Control group :( 30 participants ) will only exercise Study protocol:The randomized experimental and control group will study 3 days per week for a total of 8 weeks .Exercises difficulty;Borg Scale(0-10):It will be modarate.

Evaluation:All evaluations will be made as a Pre-test/Post-test. The detailed descriptions and characteristics of the participants will be summarized at baseline and after 8 weeks, and the differences between groups, intergroup differences will be statistically evaluated.

DETAILED DESCRIPTION:
Purpose of the research:To investigate the effects of exercises combined with action observation on balance and fall risk in individuals over 65 years of age.

The hypothesis of the research is that action observation will be more useful in maintaining balance and preventing the risk of failling.

Action observation therapy (AOT)is a novel rehabilitation technique, which involves observation of purposeful actions with the intention to imitate and then performing those actions. AOT can be described as the patient being asked to carefully observe actions presented through a video-clip or performed by an operator, in order to imitate, try, and execute them after observation .This may include the mirror neuron system (MNS) processes on the upper limb function resulting from the observation of actions (new motor skills) and actual execution of similar neural structures . Current evidence have been limited to investigating AOT effectiveness on upper and lower limb rehabilitation in both neurological and orthopedic disorders, patients with stroke and brain injuries, limb pain, Parkinson disease, and in the old women. However, despite the volume of our understanding, there is a dearth of current scientific evidence evaluating the efficacy of AOT combined with exercises on balance and risk of fall in elderly both in men and women.

Study Power Analysis:The effect size was calculated using the G Power Package Program(G Power 3.0.10) over the data of the reference article(Leem SH et al,2019).The sample size required for the study according to the calculated effect size was determined as at least 38 participants for %95 power and Type I error rate (alpha):0.05 were calculated.To increase the power of our study, we invited 100 volunteer participants and after the exclusion criteria, we started with 60 participants, but with 43 participants.We were able to complete our work.

Our research is a randomized, controlled experimental study that examines the effect of Action Observation Therapy (EGT) on balance and fall risk in individuals over the age of 65, with a probabilistic, systematic sample.

Study protocol:

Participants will be randomly divided into two groups as experimental and control groups.

Experimental group participants:(n=30) Action observation+ exercise combination Control group participants:(n=30) Only exercise A total of 43 participants completed the study as 22 participants in the experimental group and 21 participants in the control group for various reasons.

Experimental group , the participants will be asked to carefully observe actions presented through a video-clip exercise for 15 minutes, and then do same exercises for about 45 minutes in 5-10 repetitions.

The Control group (only exercise group), the participants will perform exercises for about 45 minutes in 5-10 repetitions without a video-clip observation.

Study program:3 days a week for 8 weeks Exercise difficulty:Modified Borg Scale(0-10); The modified Borg Scale was used to evaluate the intensity and difficulty grades of the exercises . Initially, the scores of 3 and 4 were applied, and a gradual increase up to 5 and 6 at the end of the studyExercise program:Exercises will be easy to learn but not complex in terms of recall and performans. Depending on the fitness of the person, %50-75 of the maximum heart rate (220-years),the exercise intensity will be preferred over the Borg Scale.

The center where the research will be conducted ,İstanbul-Beşiktaş District Abbasağa neighborhood.

Exercises;sitting and standing from easy to difficult; it will be advanced from those done with two feed touching the ground to those done on one foot and walking. It will include warm-up period, strengthening exercises ,static and dynamic balance exercises, flexibility exercises and cooling periods. The exercises were repeated 5 times initially. Then their repetition numbers were gradually increased up to 8-10 repetitions in small groups of 5-7 people.All AOT and exercise programs were performed in the Abbasağa garden park, a quiet place without noise. We obtained local permission from Besiktas Municipality, Istanbul, Turkey, and applied the general rules for the COVID-19 pandemic.The participant registration and acceptance of this study and the implementation of the exercises protocol were made by the same research physical therapist.

Study start date: December-2020

Study application date: 1 April / 31 May 2021

Completion of research: December-2021

Evaluation: All evaluations will be made as a Pre-test/ Post-test The detailed descriptions and characteristics of the participants will be summarized at baseline and after 8 weeks, and the differences between groups, intergroup differences will be statistically evaluated.

Socio-demographic evaluation Blood pressure and heart rate measurement Mini-Mental Test İnternational Physical Activity Questionnaire Short Form(IPAQ-Short)

Cognitive Level Tests :

Montreal Cognitive Assessment(MoCA)

Balance and Fall Risk Tests:

Time Up&Go Test(TUG) 5 Times Sit & Stand Test Tinetti Balance and Walk Test Activity Specific Balance Confidence Scale(ABC) BORG Scale (0-10): To determine exercise intensity I have prepared '' Pain Location and İntensity" and "Fall Frequency Questioning"and "Participant Satisfaction" evaluation forms in the last year.

Statistical evaluation: The evaluation of the all data will be done using the SPSS statistical package program.The data will be analyzed using the SPSS program with the significance level of p<0.05

İstanbul Medıpol Unıversıty Non-İnterventional Clinical Research Ethıcs Committee Permission of the research was obteined(Number:10840098-772.02-E.58328,Date:10/26/2020).

ELIGIBILITY:
Inclusion Criteria:

* Those who volunteered to participate in the study and between the ages of 65 and 80
* Who scored 24 or more out of 30 points in the Standardized Mini-Mental Test (SMMT)
* Non-neurological or orthopedic problems
* Had vision and hearing problems at a level that would prevent participation in the study.

Exclusion Criteria:

* Those who have any neurological, internal or orthopedic problems that may affect the balance,
* Those with unstable hypertension and diabetes,
* Those with a diagnosis of Chronic Obstructive Pulmonary Disease (COPD),
* Those who have had a surgical procedure that may affect the balance in the last 6 months were excluded from the study.
* Wheelchair dependents

Ages: 65 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 43 (Actual)
Dates: Start 2020-12-12 (Actual); Primary Completion 2021-04-01 (Actual); Study Completion 2021-05-31 (Actual)

PRIMARY OUTCOMES:
Mini-Mental State Examination | Baseline
  Mini Mental State Test is a short test used for dementia screening. It consists of ten questions. It measures orientation, memory, attention, calculation, language, motor function and perception, immediate and brief recall, language and simple verbal and written instructions as well as visual construction. The test is evaluated over 30 points. Between 24-30 points is considered normal and below 23 points is considered risk of dementia.This test is also affected by age and education level. The test used as the acceptance of the study participants to the research.
Baseline characteristics of the participants | Baseline
  To interpret the results of our study, baseline characteristics of the participants including age, gender, education, marital status, height, weight will be recorded.
Montreal Cognitive Assessment Scale | Baseline to end of week 8 when the study is completed.
  Montreal Cognitive Assessment Scale is a rapid screening test for measuring cognitive level and mild cognitive impairment.
  With the Montreal Cognitive Assessment Test, 8 different cognitive functions are evaluated: attention and concentration, executive functions, memory, language, visual structuring skills, abstract thinking, calculation and orientation. The highest score that can be obtained from the test is 30. Accordingly, 21 points and above is considered normal.
The International Physical Activity Questionnaire short form | Baseline.
  The short form IPAQ is a 7-item scale, assessing the amount of minutes spent in vigorous and moderate intense activity and walking during the last 7 days. For all categories, the amount of Metabolic Equivalents (METs) minutes is calculated by multiplying the amount of minutes with 8 (vigorous), 4 (moderate), 3.3 (walking), or 1.3 (sitting).
Five Times Sit-to-Stand Test | Baseline to end of week 8 when the study is completed.
  The Five Times Sit and Stand Test is a clinical test that investigates postural control and lower extremity muscle strength. It is determined by measuring the time to complete the sitting-stand up activity at least five times with a stopwatch. Completion time below 12 seconds is considered a risk for recurrent falls.
Tinetti Balance and Gait Scale | Baseline to end of week 8 when the study is completed.
  Tinetti's balance and gait scale is used to determine fall risk, especially in the elderly. It is a combination of two scales, one evaluating balance and gait characteristics. The full scale is calculated by summing the questions consisting of 9 items for balance and 7 items for walking, and evaluation scores such as 0-1-2. It is calculated by adding a maximum balance score of 16 points and a maximum walking score of 12 points. The total score is 28 as balance + walking. 18 points and below indicate high fall risk, 19-24 points medium fall risk, 24 points and above indicate low fall risk.
Activity Specific Balance Confidence Scale | Baseline to end of week 8 when the study is completed.
  Activity Specific Balance Confidence Scale was developed by Powell and Myers. This scale includes 16 tasks related to indoor and outdoor activities of daily living to balance trust in older people with varying levels of functioning. Scores range from 0 percent (no confidence) to 100 percent (complete confidence) for each question item. Higher scores with a percentage increase indicate more confidence.
Heart rate measurement | Day 1
  There are many circulatory changes that occur during exercise to supply the tremendous blood flow required by the muscles including the stimulatory effects on the circulation by the mass sympathetic discharge, the increased arterial pressure and cardiac output. These cardiovascular responses is important that adults, and elderly normal people due to the age related. It was preferred that the exercises should be percent of the maximum heart rate (220-age) according to the fitness level of the participant and the exercise difficulty level should be at the moderate.
Borg Scale assessment of perceived effort | Day 1
  Borg Scale It is the marking of the exercise intensity, which is determined by a certain percentage of the calculation of the maximum heart rate according to the fitness level of the participant, by expressing the exercise intensity in the form with numbers 1-10.The exercise difficulty is indicated by the numbers 1 through 10, with 1 being the easiest and 10 the hardest.
International Physical Activity Questionnaire Short Form | Baseline
  This is a questionnaire scale to determine the physical activity levels of the participants. This questionnaire consists of 4 parts as work, transportation, rest and sports activities. It is a 9-item scale that evaluates the amount of minutes spent for at least 10 minutes of vigorous, moderate activities and walking categories during the last 7 days. It is calculated by multiplying the minutes spent in each category by the metabolic equivalent. Under the 600 metabolic equivalents are considered inactive, 600-3000 metabolic equivalents minimum active and 3000 metabolic equivalents as active.
The Timed Up and Go Test | Baseline to end of week 8 when the study is completed.
  In balance and fall risk assessments, the Timed Get Up and Go Test (TUGT) is a simple and very useful test.A chair and stopwatch are required for this test.The area of 3 meters in front of the chair is determined. The patient is asked to get up from the chair and walk this distance and sit down again.If an elderly individual completes this test in more than 12 seconds, there is a risk of falling

SECONDARY OUTCOMES:
The frequency of falling | Baseline
  The frequency of falling will be determined by self questioning
Clinical pain location and pain intensity | Baseline to end of week 8 when the study is completed.
  In this test to determine the participant's clinical pain location and the severity of that pain. The participant is asked to mark the area of pain on the form with a human body template. Pain severity, which is also in the same form, is evaluated on a scale of 0-10 points. Zero means "no pain" and 10 means "pain as bad as possible".

OTHER OUTCOMES:
Research Participant Satisfaction Questionnaire | At the end of the 8th week of completion.
  In the questionnaire, we ask questions about the informed consent process, interaction with the research team, satisfaction with the study, and how easy it is to complete the study. Higher scores mean higher satisfaction

CONTACTS AND LOCATIONS:
Overall Officials: Bağdat TEKKUŞ, 1, Principal Investigator — Istanbul MEDİPOL University ,İnstitute of Health Sciences Kavacık Campus-İstanbul TURKEY; Fatma MUTLUAY, 2, Study Director — Istanbul MEDİPOL University Faculty of Health Sciences Professor
Locations (1):
- Istanbul Medipol University Kavacık Campus, Istanbul, Kavacık, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
I can consider publishing my research as a doctoral thesis and related article.

REFERENCES:
- [Background] Leem SH, Kim JH, Lee BH. Effects of Otago exercise combined with action observation training on balance and gait in the old people. J Exerc Rehabil. 2019 Dec 31;15(6):848-854. doi: 10.12965/jer.1938720.360. eCollection 2019 Dec. PMID 31938708
- [Background] Gangitano M, Mottaghy FM, Pascual-Leone A. Phase-specific modulation of cortical motor output during movement observation. Neuroreport. 2001 May 25;12(7):1489-92. doi: 10.1097/00001756-200105250-00038. PMID 11388435
- [Background] Bird ML, Hill K, Ball M, Williams AD. Effects of resistance- and flexibility-exercise interventions on balance and related measures in older adults. J Aging Phys Act. 2009 Oct;17(4):444-54. doi: 10.1123/japa.17.4.444. PMID 19940323
- [Background] Martins AC, Santos C, Silva C, Baltazar D, Moreira J, Tavares N. Does modified Otago Exercise Program improves balance in older people? A systematic review. Prev Med Rep. 2018 Jul 10;11:231-239. doi: 10.1016/j.pmedr.2018.06.015. eCollection 2018 Sep. PMID 30210995
- [Background] Gatti R, Sarasso E, Pelachin M, Agosta F, Filippi M, Tettamanti A. Can action observation modulate balance performance in healthy subjects? Arch Physiother. 2019 Jan 22;9:1. doi: 10.1186/s40945-018-0053-0. eCollection 2019. PMID 30693101
- [Background] Hirvensalo M, Heikkinen E, Lintunen T, Rantanen T. Recommendations for and warnings against physical activity given to older people by health care professionals. Prev Med. 2005 Jul;41(1):342-7. doi: 10.1016/j.ypmed.2004.11.020. PMID 15917031
- [Background] Parry SW, Finch T, Deary V. How should we manage fear of falling in older adults living in the community? BMJ. 2013 May 28;346:f2933. doi: 10.1136/bmj.f2933. No abstract available. PMID 23714190
- [Background] Sherrington C, Tiedemann A, Fairhall N, Close JC, Lord SR. Exercise to prevent falls in older adults: an updated meta-analysis and best practice recommendations. N S W Public Health Bull. 2011 Jun;22(3-4):78-83. doi: 10.1071/NB10056. PMID 21632004
- [Background] Pelosin E, Barella R, Bet C, Magioncalda E, Putzolu M, Di Biasio F, Cerulli C, Casaleggio M, Abbruzzese G, Avanzino L. Effect of Group-Based Rehabilitation Combining Action Observation with Physiotherapy on Freezing of Gait in Parkinson's Disease. Neural Plast. 2018 May 27;2018:4897276. doi: 10.1155/2018/4897276. eCollection 2018. PMID 29977280
- [Background] Buccino G. Action observation treatment: a novel tool in neurorehabilitation. Philos Trans R Soc Lond B Biol Sci. 2014 Apr 28;369(1644):20130185. doi: 10.1098/rstb.2013.0185. Print 2014. PMID 24778380
- [Background] Caligiore D, Mustile M, Spalletta G, Baldassarre G. Action observation and motor imagery for rehabilitation in Parkinson's disease: A systematic review and an integrative hypothesis. Neurosci Biobehav Rev. 2017 Jan;72:210-222. doi: 10.1016/j.neubiorev.2016.11.005. Epub 2016 Nov 16. PMID 27865800
- [Background] Villafane JH, Pirali C, Isgro M, Vanti C, Buraschi R, Negrini S. Effects of Action Observation Therapy in Patients Recovering From Total Hip Arthroplasty Arthroplasty: A Prospective Clinical Trial. J Chiropr Med. 2016 Dec;15(4):229-234. doi: 10.1016/j.jcm.2016.08.011. Epub 2016 Oct 5. PMID 27857630
- [Background] Zhu MH, Wang J, Gu XD, Shi MF, Zeng M, Wang CY, Chen QY, Fu JM. Effect of action observation therapy on daily activities and motor recovery in stroke patients.International Journal of Nursing Sciences. 2015 Sep 1;2(3):279-82.
- [Background] Gardner MM, Buchner DM, Robertson MC, Campbell AJ. Practical implementation of an exercise-based falls prevention programme. Age Ageing. 2001 Jan;30(1):77-83. doi: 10.1093/ageing/30.1.77. PMID 11322678
- [Background] Çifcili S,Ünalan P.Yaşlılarda fonksiyonel kayıplara yaklaşım.Turk Aile Hek Dergisi 2004;8:166-173.
- [Background] World Health Organisation (WHO) Falls. 2018.
- [Background] Alamer A, Melese H, Adugna B. Effectiveness of Action Observation Training on Upper Limb Motor Function in Children with Hemiplegic Cerebral Palsy: A Systematic Review of Randomized Controlled Trials. Pediatric Health Med Ther. 2020 Sep 15;11:335-346. doi: 10.2147/PHMT.S266720. eCollection 2020. PMID 32982541
- [Background] Zhu M-H, Wang J, Gu X-D, et al. Effect of action observation therapy on daily activities and motor recovery in stroke patients. Int J Nurs Stud. 2015;2(3):279-282. doi:10.1016/j.ijnss.2015.08.006
- [Background] Buccino G, Binkofski F, Fink GR, Fadiga L, Fogassi L, Gallese V, Seitz RJ, Zilles K, Rizzolatti G, Freund HJ. Action observation activates premotor and parietal areas in a somatotopic manner: an fMRI study. Eur J Neurosci. 2001 Jan;13(2):400-4. PMID 11168545
- [Background] Dinomais M, Lignon G, Chinier E, Richard I, Ter Minassian A, Tich SN. Effect of observation of simple hand movement on brain activations in patients with unilateral cerebral palsy: an fMRI study. Res Dev Disabil. 2013 Jun;34(6):1928-37. doi: 10.1016/j.ridd.2013.03.020. Epub 2013 Apr 11. PMID 23584173
- [Background] Rizzolatti G, Fadiga L, Gallese V, Fogassi L. Premotor cortex and the recognition of motor actions. Brain Res Cogn Brain Res. 1996 Mar;3(2):131-41. doi: 10.1016/0926-6410(95)00038-0. PMID 8713554
- [Background] Sgandurra G, Biagi L, Fogassi L, Sicola E, Ferrari A, Guzzetta A, Tosetti M, Cioni G. Reorganization of the Action Observation Network and Sensory-Motor System in Children with Unilateral Cerebral Palsy: An fMRI Study. Neural Plast. 2018 Jul 25;2018:6950547. doi: 10.1155/2018/6950547. eCollection 2018. PMID 30147718
- [Background] Sarasso E, Gemma M, Agosta F, Filippi M, Gatti R. Action observation training to improve motor function recovery: a systematic review. Arch Physiother. 2015 Dec 2;5:14. doi: 10.1186/s40945-015-0013-x. eCollection 2015. PMID 29340183
- [Background] Borges LR, Fernandes AB, Melo LP, Guerra RO, Campos TF. Action observation for upper limb rehabilitation after stroke. Cochrane Database Syst Rev. 2018 Oct 31;10(10):CD011887. doi: 10.1002/14651858.CD011887.pub2. PMID 30380586
- [Background] Buchignani B, Beani E, Pomeroy V, Iacono O, Sicola E, Perazza S, Bieber E, Feys H, Klingels K, Cioni G, Sgandurra G. Action observation training for rehabilitation in brain injuries: a systematic review and meta-analysis. BMC Neurol. 2019 Dec 27;19(1):344. doi: 10.1186/s12883-019-1533-x. PMID 31881854
- [Background] Peng TH, Zhu JD, Chen CC, Tai RY, Lee CY, Hsieh YW. Action observation therapy for improving arm function, walking ability, and daily activity performance after stroke: a systematic review and meta-analysis. Clin Rehabil. 2019 Aug;33(8):1277-1285. doi: 10.1177/0269215519839108. Epub 2019 Apr 12. PMID 30977387
- [Background] Thieme H, Morkisch N, Rietz C, Dohle C, Borgetto B. The Efficacy of Movement Representation Techniques for Treatment of Limb Pain--A Systematic Review and Meta-Analysis. J Pain. 2016 Feb;17(2):167-80. doi: 10.1016/j.jpain.2015.10.015. Epub 2015 Nov 6. PMID 26552501
- [Background] Meeus M, Van Eupen I, Willems J, Kos D, Nijs J. Is the International Physical Activity Questionnaire-short form (IPAQ-SF) valid for assessing physical activity in Chronic Fatigue Syndrome? Disabil Rehabil. 2011;33(1):9-16. doi: 10.3109/09638288.2010.483307. Epub 2010 May 6. PMID 20446802
- [Background] Cumming TB, Bernhardt J, Linden T. The montreal cognitive assessment: short cognitive evaluation in a large stroke trial. Stroke. 2011 Sep;42(9):2642-4. doi: 10.1161/STROKEAHA.111.619486. Epub 2011 Jul 14. PMID 21757673
- [Background] Wallmann HW, Evans NS, Day C, Neelly KR. Interrater Reliability of the Five-Times-Sit-to-Stand Test. Home Health Care Management & Practice. 2013;25(1):13-17. doi:10.1177/1084822312453047
- [Background] Gomes Gde C, Teixeira-Salmela LF, Fonseca BE, Freitas FA, Fonseca ML, Pacheco BD, Goncalves MR, Caramelli P. Age and education influence the performance of elderly women on the dual-task Timed Up and Go test. Arq Neuropsiquiatr. 2015 Mar;73(3):187-93. doi: 10.1590/0004-282X20140233. PMID 25807122
- [Background] Souza Melo R de, Silva PWA, Tassitano RM, Macky CFST, Silva LVC. Balance and gait evaluation: comparative study between deaf and hearing students. Rev Paul Pediatr 2012; 30 (3): 385-91.
- [Background] Ayhan C, Buyukturan O, Kirdi N, Yakut Y, Guler C. The Turkish version of the activities specific balance confidence (ABC) scale: its cultural adaptation, validation and reliability in older adults. Turkish Journal of Geriatrics. 2014; 17 (2): 157-163.
- [Background] Milot MH, Leonard G, Corriveau H, Desrosiers J. Using the Borg rating of perceived exertion scale to grade the intensity of a functional training program of the affected upper limb after a stroke: a feasibility study. Clin Interv Aging. 2018 Dec 19;14:9-16. doi: 10.2147/CIA.S179691. eCollection 2019. PMID 30587949
- [Background] Sjahris H, Ritarwan K, Tarigan S, Rambe AS, Lubis ID, Bhakti I. The mini mental state examination in healthy individuals in Medan, Indonesia by age and education level. Neurol J Southest Asia. 2001; 6: 19-22.
- [Background] Hassan AE. Heart Rate and Blood Pressure Responses to Exercise Testing in Relation to Age in Healthy Men. The Iraqi Postgraduate Medical Journal. 2009; 1(1): 14-20.
- [Derived] Drahota A, Udell JE, Mackenzie H, Pugh MT. Psychological and educational interventions for preventing falls in older people living in the community. Cochrane Database Syst Rev. 2024 Oct 3;10(10):CD013480. doi: 10.1002/14651858.CD013480.pub2. PMID 39360568
- [Derived] Tekkus B, Mutluay F. Effect of community-based group exercises combined with action observation on physical and cognitive performance in older adults during the Covid-19 pandemic: A randomized controlled trial. PLoS One. 2023 Dec 5;18(12):e0295057. doi: 10.1371/journal.pone.0295057. eCollection 2023. PMID 38051723